CLINICAL TRIAL: NCT05529069
Title: Phase II Study of Pirtobrutinib With Venetoclax In Relapsed-Refractory MCL (Mantle Cell Lymphoma) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Loxo Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1108; NCI-2022-07498 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Mantle Cell Lymphoma; Non Hodgkin Lymphoma; Hematologic Malignancy
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Hematologic Neoplasms | interventions — pirtobrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pirtobrutinib (LOXO-305) and Venetoclax (combination) (Experimental): Participants will have study visits every week during Cycle 1, and then on Day 1 of every cycle for the first year. After that, they will have study visits on Day 1 of every 2 cycles.
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Pirtobrutinib — Given by PO
  Other Names: LOXO-305
Drug: Venetoclax — Given by PO
  Other Names: ABT-199,

SUMMARY:
To learn if the combination of pirtobrutinib (also called LOXO-305) and venetoclax can help to control mantle cell lymphoma (MCL) that is relapsed (has come back) or refractory (has not responded to therapy).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

• To determine the efficacy (overall response rate) and safety profile of the Pirtobrutinib plus venetoclax combination in relapsed refractory MCL patients

SECONDARY OBJECTIVE:

• To evaluate the survival (including overall and progression-free survival) of the Pirtobrutinib plus venetoclax combination in relapsed refractory MCL patients.

EXPLORATORY STUDIES:

•Exploratory studies are planned on the trial and the final analysis and methodology including bio-informatics analysis

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of mantle cell lymphoma in tissue biopsy by hematopathology with/without chromosome translocation t(11;14), (q13;q32) and/or overexpress cyclin D1 in tissue biopsy. Cyclin D1 negative MCL (confirmed by hematopathology at MDACC are allowed).
2. The patient is able to take oral medications
3. Relapsed MCL (irrespective of prognostic factors) including any lines or prior therapy or patients who had prior ibrutinib, acalabrutinib, zanubrutinib, other BTK inhibitor or anti CD19-CART therapy, single agent or in combination (without prior venetoclax) or relapsed high risk MCL including any or all of the following (Blastoid/pleomorphic histology), High Ki-67 (≥50%), TP53 mutated or del17p by FISH, NSD2, NOTCH2, CDKN2A mutated or MYC positive by FISH or MYC, Bcl2 amplification, complex karyotype or high risk biologic MIPI score
4. Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
5. Age from >=18 years at the time of signing the informed consent.
6. Patients may have at least 1 site of radiographically assessable disease (i.e., lymph node longest diameter [LDi] >= 1.5 cm, not necessary for disease assessable by positron emission tomography [PET]/computerized tomography [CT], extra nodal site >= 1.0 cm in LDi. Patients with BM only or GI only relapse are allowed.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.
8. Disease free of prior malignancies with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or other malignancies in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years pertaining to prior malignancy. PI could use judgment in the best interest of patients.
9. Patients must have relapsed or refractory MCL (irrespective of prior BTK inhibitor or anti CD19 CART exposure).
10. Prothrombin time (or international normalized ratio) and partial thromboplastin time not to exceed 1.2 times the institutional upper limit of normal range (patients with an elevated prothrombin time and known lupus anticoagulant may be eligible for participation after consulting the IND sponsor).
11. Adequate BM function independent of growth factor or PRBC or platelet transfusion support (within 14 days of Screening assessment and criteria must be met on C1D1 without transfusion/G-CSF within 7 days of assessment, per local laboratory reference range at screening as follows:

    1. platelet count >=50, 000/mm3;
    2. absolute neutrophil count (ANC) >= 1000/mm3 unless cytopenia is clearly due to marrow involvement from MCL
    3. total hemoglobin >= 8 g/dL (without transfusion support within 2 weeks of screening); If any of the above-mentioned cytopenias (a-c) are present due to significant BM involvement, at least 30% BM involvement by MCL (requiring transfusion or granulocyte colony-stimulating factor [G-CSF] support) MCL patients may proceed with enrollment after discussion with the PI or Co-PI. Cytopenias may not be due to evidence of myelodysplastic syndrome (MDS) or hypoplastic BM.
12. Adequate organ function as defined by the following laboratory values:

    1. Creatinine clearance. >=30 mL/min (by Cockcroft-Gault method, APPENDIX I),
    2. Total bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN with documented liver involvement and/or Gilbert's Disease or controlled immune hemolysis or considered an effect of regular blood transfusions.
    3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 x ULN, or < 5 x upper limit of normal if hepatic metastases are present.
13. Projected life expectancy of >12 weeks pertaining to lymphoma.
14. Female patients must be surgically sterile, postmenopausal (for at least 1 year), or have confirmed negative results for a pregnancy test at screening, on a blood or urine sample obtained within 7 days prior to initiation of study treatment.
15. Women of childbearing potential and men with female partners of childbearing potential must be willing to use an effective form of contraception for at least 6 months after the last dose of study treatment. Patient enrolled into the Pirtobrutinib+ venetoclax study should use an effective form of contraception for 6 months after the last dose of Pirtobrutinib in combination with venetoclax, whichever time period is longer. Recommended methods of highly effective birth control are:

    * Hormonal contraception (birth control pills, patches, or rings)
    * Intrauterine device (IUD)
    * Birth control injections
    * Double barrier methods (diaphragm with spermicidal gel or condoms with birth control foam)
    * Sterilization of participant or partner ("tubes tied" or vasectomy) Willingness of men and women of reproductive potential (defined as following menarche and not postmenopausal [and 2 years of non-therapy-induced amenorrhea] or surgically sterile) to observe conventional and highly effective birth control methods with failure rates of < 1% for the duration of treatment and for 6 months following the last dose of study treatment; this must include barrier methods such as condom or diaphragm with spermicidal gel. Women of reproductive potential are defined as following menarche and not postmenopausal (and 2 years of non-therapy-induced amenorrhea) or surgically sterile. For male subjects with a non-pregnant female partner of child-bearing potential and a woman of child-bearing potential one of the following highly effective birth control methods with a failure rate of less than 1% per year when used consistently and correctly are recommended: Combined estrogen and progestin containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or trans dermally, progestin-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant, Intrauterine device (IUD) , Intrauterine hormone-releasing system (IUS), Bilateral tubal occlusion, Vasectomized partner, Sexual abstinence: considered a highly effective method only if defined as refraining from heterosexual intercourse during an entire period of risk associated with the study treatment. The reliability of sexual abstinence will be evaluated in relation to the duration of the study and to the usual lifestyle of the subject (CTFG 2014).

    Birth control methods unacceptable for this clinical trial are:
    1. Periodic abstinence (calendar, hypothermal, or post-ovulation methods)
    2. Withdrawal (coitus interruptus)
    3. Spermicide only
    4. Lactational amenorrhea method • Sperm donation is prohibited during the duration of participation on this protocol and for 6 months after the last dose of any study drug.
16. Patients are required to have the following washout periods prior to planned Cycle 1 Day 1 (C1D1).

    * Targeted agents, investigational agents, therapeutic monoclonal antibodies or cytotoxic chemotherapy: 5 half-lives or 2 weeks, whichever is shorter
    * Immunoconjugates antibody treatment within 10 weeks prior to enrollment.
    * Broad field radiation (≥ 30% of the bone marrow or whole brain radiotherapy) must be completed 28 days prior to study enrollment
    * Palliative limited field radiation must be completed 7 days prior to study enrollment. Note: In the case of known central nervous system (CNS) involvement by systemic lymphoma: Patients with previous treatment for CNS involvement who are neurologically stable and without evidence of disease may be eligible if a compelling clinical rationale is provided by the Investigator and with documented IND sponsor's approval.
17. Prior treatment-related AEs must have recovered to Grade ≤ 1 with the exception of alopecia and Grade 2 peripheral neuropathy.

Exclusion Criteria:

1. Known central nervous system (CNS) involvement by lymphoma. Patients with previous treatment for CNS involvement who are neurologically stable and without evidence of disease (as shown by MRI brain and/or CSF or clinical exam by neurologists may be eligible if a compelling clinical rationale is provided to institutional IND sponsor contact.)
2. History of bleeding diathesis
3. History of stroke or intracranial hemorrhage within 6 months of C1D1
4. Vaccination with live vaccine within 28 days prior to enrollment.
5. Have a known hypersensitivity to any of the excipients of Pirtobrutinib or to the intended covalent BTK inhibitor if randomized to control arm.
6. Patients who experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor. NOTE: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome).
7. Pregnant or lactating females.
8. Known and uncontrolled HIV infection. Participants with HIV (known HIV 1/2 antibodies positive) are allowed if all of the following conditions are met:

   * CD4+ T-cell counts ≥350 cells/μL;
   * Participants with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections may be eligible, if they have not had an opportunistic infection within the past 12 months;
   * If participant is on antiretroviral, evaluation of the specific agents must be performed in order to determine if participant is eligible (e.g., excluding patients taking strong CYP3A inhibitors such as ritonavir). If necessary, evaluate the feasibility of switching to an alternate effective ARV therapy (ART) regimen before study participation. Participants need to be on established ART for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
   * Screening for HIV infection is not required
9. Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below: Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before enrollment. Patients who are hepatitis B PCR positive will be excluded. Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before enrollment. Patients who are hepatitis C RNA positive will be excluded.
10. Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator and IND sponsor may pose a risk for patient participation. Screening for chronic conditions is not required.
11. Pregnancy, lactation or plan to breastfeed during the study or within 6 months of the last dose of study treatment
12. Significant cardiovascular disease defined as:

    * unstable angina or acute coronary syndrome within the past 2 months prior to enrollment
    * history of myocardial infarction within 3 months prior to enrollment or
    * documented LVEF by any method of ≤ 40% in the 12 months prior to enrollment
    * ≥ Grade 3 NYHA functional classification system of heart failure, uncontrolled or symptomatic arrhythmias
13. Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec on at least 2/3 consecutive electrocardiograms (ECGs), and mean QTcF > 470 msec on ECG, during Screening. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33).

    * Correction of suspected drug induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
    * Correction for underlying bundle branch block (BBB) allowed. Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker.
14. Concomitant malignancies or previous malignancies with less than a 1-year disease-free interval at the time of signing consent. Subjects with adequately treated basal or squamous cell carcinoma of the skin, or adequately treated carcinoma in situ (e.g. cervix) may enroll irrespective of the time of diagnosis. Patients with controlled, advanced prostate cancer (not on active chemotherapy) are permitted. Active second malignancy unless in remission with life expectancy > 2 years. Examples include:

    * a. Adequately treated no melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease.
    * b. Adequately treated cervical carcinoma in situ without current evidence of disease.
    * c. Localized (e.g., lymph node negative) breast cancer treated with curative intent with no evidence of active disease present for more than 3 years and receiving adjuvant hormonal therapy.
    * d. Localized prostate cancer undergoing active surveillance.
15. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of venetoclax.
16. With known allergies to xanthine oxidase inhibitors and/or rasburicase.
17. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study.
18. No concomitant anticancer therapies, immunotherapies, cellular, or radiotherapy. No major surgery within 4 weeks prior to first dose of study treatment. Washout period for chemotherapy is 14 days. Washout period for targeted agents is 2 weeks or 5 half-lives (t1/2) (whichever is shorter). Washout period for antibody-based immunotherapies or cellular therapies is 4 weeks. Washout period for radiotherapy is 7 days (limited field) and 28 days (extended field that includes BM). Washout period must be completed prior to any treatment administration.
19. Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenia. Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) is for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts.
20. Concomitant steroids for disease related pain control are allowed at any dose but must be discontinued prior to any study treatment initiation. Chronic use of corticosteroids is allowed up to 20 mg prednisone or equivalent daily for non-cancer related conditions at the time of study start.
21. History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T cell (CAR-T) therapy within 60 days of enrollment or presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing: • active graft versus host disease (GVHD); • cytopenia from incomplete blood cell count recovery post-transplant; • need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy; • ongoing immunosuppressive therapy (> 20 mg prednisone or equivalent daily).
22. Known neurologic disorder or residual neurologic toxicities that may put patients at increased risk of neurologic toxicity in the opinion of the investigator.
23. Active uncontrolled systemic infection.
24. Received an investigational agent within 2 weeks or within 5 T1/2, whichever is shorter prior to the first dose of study treatment.
25. Current treatment with certain strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and/or strong P-gp inhibitors. Because of their effect on CYP3A4, use of any of the following within 3 days of study therapy start or planned use during study participation is prohibited, • grapefruit or grapefruit products

    * Seville oranges or products from Seville oranges
    * star fruit
26. Patients taking warfarin and/or equivalent vitamin K antagonists are excluded since the use of these agents is contraindicated with Pirtobrutinib or with venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
ORR (overall response rate) | through study completion an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Preetesh Jain, MD, DM, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://mdanderson.org